CLINICAL TRIAL: NCT00400257
Title: SCREEN-HF (Screening Evaluation of the Evolution of New Heart Failure)
Brief Title: Screening Evaluation of the Evolution of New Heart Failure (SCREEN-HF)
Status: Completed | Type: Observational
Sponsor: Ingrid Hopper (Other)
Collaborators: HBA (Unknown)
Responsible Party: Sponsor-Investigator, Ingrid Hopper, Dr Ingrid Hopper, The Alfred
Organization: The Alfred (Other)
Other Study IDs: CP-04/06
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; BNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: People at high risk of heart failure.
  Interventions: Behavioral: Early detection of heart failure

INTERVENTIONS:
Behavioral: Early detection of heart failure — Early detection of heart failure

SUMMARY:
The investigators are hoping to identify early heart failure in patients who do not have symptoms as yet and at the same time assess the usefulness of Brain natriuretic peptide (BNP) in doing this.

DETAILED DESCRIPTION:
Measuring Brain natriuretic peptide (BNP) and N-terminal proBNP (NT-proBNP)and can give us useful information about a persons heart function in patients with symptoms such as shortness of breath. This is because BNP/NT-proBNP levels rise when the heart is under pressure as it is in people with heart disease. However, we don't know if this is a useful test to do in people who are at a high risk of developing heart disease but who have no symptoms and have not been diagnosed with any heart problems.

In this study we hope to recruit 3500 participants. This study is being run in conjunction with HBA (recently renamed Bupa) and we estimate that 10,000 HBA members will need to be contacted by letter and invited to screen for this study to achieve the required 3500 (protocol amended to include people who meet the entry criteria but who are not insured through HBA).

This protocol has been amended to allow us to invite 50 participants with the lowest NT-proBNP levels to also continue in the study and have blood tests, an ECG and echocardiography as described below.

Participants will undergo a routine blood test which will include measuring NT-proBNP. Only participants in whom NT-proBNP is elevated will undergo additional blood tests (for cardiac markers), an ECG and echocardiography to determine if there is any indication that they do have heart disease even though they have not been diagnosed and are not symptomatic.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years
2. Have been insured with HBA for 12 months or longer (Protocol amended to remove this criteria and allow enrollment of the general public)
3. Subjects at high-risk of subsequent development of heart failure; comprising at least one of:

   * Prior myocardial infarction (MI) without known left ventricular (LV) dysfunction
   * Current active ischemic heart disease
   * Prior Cerebrovascular Accident (CVA)
   * Known valvular heart disease without known LV dysfunction
   * Atrial fibrillation
   * Ventricular arrhythmia resulting in syncope or pre-syncope (protocol amended to remove this entry criteria)
   * Treated hypertension, of at least 2 years duration
   * Treated Diabetes mellitus, of at least 2 years duration
   * Estimated Glomerular Filtration Rate (eGFR) <50ml/min

Exclusion Criteria:

1. Known systolic or diastolic heart failure
2. Symptoms suggestive of current heart failure. (protocol amended to remove this criteria)
3. LV systolic or diastolic dysfunction on echocardiography or other objective imaging modality.
4. Medications for treatment of heart failure such as ACE inhibitors, angiotensin receptor blockers (ARBs), beta-blockers or aldosterone antagonists. Use of such medications for approved indications such as hypertension, post-MI management (without known LV dysfunction) or for diabetic nephropathy is permitted. (protocol amended to remove this criteria)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People at high risk of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of BNP in determining Heart Failure in people not previously diagnosed with the condition. | at visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, Professor, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Campbell DJ, Coller JM, Gong FF, McGrady M, Boffa U, Shiel L, Liew D, Stewart S, Owen AJ, Krum H, Reid CM, Prior DL. Kidney age - chronological age difference (KCD) score provides an age-adapted measure of kidney function. BMC Nephrol. 2021 Apr 26;22(1):152. doi: 10.1186/s12882-021-02324-y. PMID 33902478
- [Derived] Gong FF, Jelinek MV, Castro JM, Coller JM, McGrady M, Boffa U, Shiel L, Liew D, Wolfe R, Stewart S, Owen AJ, Krum H, Reid CM, Prior DL, Campbell DJ. Risk factors for incident heart failure with preserved or reduced ejection fraction, and valvular heart failure, in a community-based cohort. Open Heart. 2018 Jul 23;5(2):e000782. doi: 10.1136/openhrt-2018-000782. eCollection 2018. PMID 30057766